CLINICAL TRIAL: NCT02738606
Title: Randomized Controlled Phase II Trial of Liver Resection Versus No Surgery in Patients With Liver and Unresectable Pulmonary Metastases From Colorectal Cancer
Brief Title: Liver Surgery and Chemotherapy in Treating Patients With Colorectal Cancer With Liver Metastases That Can Be Removed by Surgery and Lung Metastases That Cannot Be Removed by Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: < 75% participation
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-1133; NCI-2016-00740 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-1133 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-04-12; First posted 2016-04-14 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Colorectal Carcinoma; Metastatic Malignant Neoplasm in the Liver; Metastatic Malignant Neoplasm in the Lung; Recurrent Colorectal Carcinoma; Resectable Colorectal Carcinoma; Stage IV Colorectal Cancer AJCC v7; Stage IVA Colorectal Cancer AJCC v7; Stage IVB Colorectal Cancer AJCC v7
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Drug Therapy; Metastasectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (surgery, chemotherapy) (Experimental): Patients undergo hepatectomy and receive chemotherapy at the discretion of treating oncologist. Patients whose lung tumors become able to be removed by surgery with chemotherapy may undergo lung metastasectomy.
  Interventions: Drug: Chemotherapy; Other: Laboratory Biomarker Analysis; Procedure: Metastasectomy; Other: Quality-of-Life Assessment; Procedure: Therapeutic Conventional Surgery
- Group II (chemotherapy) (Active Comparator): Patients receive chemotherapy at the discretion of the treating oncologist. Patients whose lung tumors become able to be removed by surgery with chemotherapy may undergo lung metastasectomy.
  Interventions: Drug: Chemotherapy; Other: Laboratory Biomarker Analysis; Procedure: Metastasectomy; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Chemotherapy
  Other Names: Chemo; Chemotherapy (NOS); Chemotherapy, Cancer, General
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Metastasectomy — Undergo lung metastasectomy
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Procedure: Therapeutic Conventional Surgery — Undergo hepatectomy
  Arms: Group I (surgery, chemotherapy)

SUMMARY:
This randomized phase II trial studies how well liver surgery and chemotherapy compared to chemotherapy alone work in treating patients with colorectal cancer that has spread to the liver (liver metastases) that can be removed by surgery and that has spread to the lungs (lung metastases) that cannot be removed by surgery. Liver surgery removes a portion of the liver affected by the tumor. Chemotherapy drugs work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Liver surgery and chemotherapy may work better than chemotherapy alone in treating patients with colorectal cancer which has spread to the liver and lungs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine a survival benefit of liver resection in patients with resectable liver and unresectable low-volume pulmonary metastases from colorectal cancer.

SECONDARY OBJECTIVES:

I. To identify biomarkers in blood and resected liver specimens that correlate with survival, and development of extrahepatic and extrapulmonary metastases.

II. To assess patients' quality-of-life in each treatment arm with serial questionnaires.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients undergo hepatectomy and receive chemotherapy at the discretion of treating oncologist. Patients whose lung tumors become able to be removed by surgery with chemotherapy may undergo lung metastasectomy.

GROUP II: Patients receive chemotherapy at the discretion of the treating oncologist. Patients whose lung tumors become able to be removed by surgery with chemotherapy may undergo lung metastasectomy.

Patients are followed up every 3-6 months up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with synchronous or metachronous diagnosis of resectable liver metastases by computed tomography (CT) or magnetic resonance imaging (MRI) of the abdomen

  * Patients requiring percutaneous or intraoperative ablation of liver metastases < 2 cm in size are eligible
  * Patients who underwent prior liver resection or ablation for colorectal liver metastases are eligible
* Patients previously treated with systemic chemotherapy and/or biologic agents for colorectal cancer are eligible
* The primary tumor in the colon or rectum may be intact or resected
* Low-volume lung metastases are defined as solid pulmonary nodules < 2 cm with non-spiculated contours, no benign-appearing calcifications, and =< 14 in number, diagnosed by computed tomography of the chest or positron emission tomography (PET)
* Lung metastases will be unresectable due to anatomic location, distribution, or patients' comorbidities, as determined by review of imaging by a faculty member in the Department of Thoracic & Cardiovascular Surgery
* Patients must sign a study-specific consent form
* Patients will undergo CT imaging of the chest, abdomen, and pelvis to evaluate lung and liver metastases within 60 days of registration; for patients who cannot tolerate CT contrast or have hepatic steatosis that reduces the sensitivity of CT, MRI of the liver will be performed

Exclusion Criteria:

* Radiographic evidence of disease other than liver and lungs, with the exception of mediastinal lymph nodes < 2 cm and hepatoduodenal ligament lymphadenopathy, diagnosed by computed tomography, magnetic resonance imaging, or positron emission tomography
* Serum bilirubin >= 2 mg/dL
* Platelet count < 50,000/uL
* Eastern Cooperative Oncology Group (ECOG) performance status of 3-4
* Patient refusal to participate in randomization
* Pregnant women are excluded from this study
* Planned stereotactic body radiation therapy (SBRT) for the pulmonary metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-05-25 (Actual); Primary Completion 2025-12-05 (Actual); Study Completion 2025-12-05 (Actual)

PRIMARY OUTCOMES:
Overall survival | From the date of randomization to the date of death or the date of last follow-up, assessed up to 3 years
  The primary analysis will be performed in an intention-to-treat data set. Stratified log-rank test adjusting for the study stratification factors will be used to compare overall survival between the two treatment arms. The hazards ratio of overall survival for the surgery arm compared to the non-surgery arm will be estimated by fitting Cox proportional hazards regression models, adjusting for the effects of covariates including stratification factors.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 3 years
  Tabulated by frequency and percentages, by grade, and by their relations to surgical treatment.
Extrahepatic and extrapulmonary metastases | Up to 3 years
  The Kaplan-Meier method will be used to estimate time to extrahepatic and extrapulmonary metastases.
Intrahepatic recurrence | Up to 3 years
  The Kaplan-Meier method will be used to estimate time to intrahepatic recurrence among patients randomized to surgery.
Biomarker levels in blood and resected liver specimens | Up to 3 years
  Univariate and multivariate Cox proportional hazards models will be fitted to evaluate the association between biomarkers in blood and resected liver specimens and time to event outcomes, including overall survival development of extrahepatic and extrapulmonary metastases, and time to intrahepatic recurrence among patients randomized to surgery. Univariate and multivariate logistic regression will be used to assess the association between biomarkers and response to chemotherapy
Scores of the Functional Assessment of Cancer Therapy - General 7 questionnaire | Up to 3 years
  Summarized using descriptive statistics including mean, standard deviation, median, and range. Summation of item GP1, GP4, GP2, and GE6 (higher score indicates worse condition) and summation of GF5, GF3 and GF7 (higher score indicates better condition) will be calculated for each patient. Two sample t-tests will be used to compare scores of each item or summations between the two treatment arms.
Patients who abandon treatment | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Yun S Chun, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/06/NCT02738606/ICF_000.pdf